CLINICAL TRIAL: NCT01253798
Title: What Type of Group Exercise Should be Chosen for Osteoarthritis Patients in the Rehabilitation Phase Following Hip Replacement Surgery?
Brief Title: Group Exercise After Hip Replacement Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitement unsuccessful
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTNU-ISM-KH-2010
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis, Hip
Keywords: exercise; hydrotherapy
MeSH Terms: conditions — Osteoarthritis, Hip; Motor Activity | interventions — Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group training on land (Active Comparator): Group training in water and on land are carried out by the same principles, which is to improve general function, and to improve function and strength around the operated hip.
  Interventions: Other: Group training
- Group training in water (Active Comparator): Group training in water and on land are carried out by the same principles, which is to improve general function, and to improve function and strength around the operated hip
  Interventions: Other: Group training

INTERVENTIONS:
Other: Group training — Each session lasts 50 minutes and consists of warm-up, mobility training, strength training, balance training and endurance training. Mobility training is conducted to increase range of motion in the operated hip, strength exercises are conducted to strengthen muscles around the operated hip, balance training are conducted to improve stability around the operated hip and endurance training are conducted to increase patients' physical capacity. This is in line with current guidelines for the exercise of osteoarthritis patients.

SUMMARY:
The purpose of this study is to determine which group exercise one should choose when hip osteoarthritis patients have undergone hip replacement surgery. To determine this, we want to answer the following research question:

Are there differences in function and muscle strength in osteoarthritis patients who conduct group training either on land or in water in the rehabilitation phase following hip replacement surgery?

ELIGIBILITY:
Inclusion Criteria:

* Hip osteoarthritis patients who undergo surgery with total prosthesis at St. Olav's Hospital, Department Orkdal.
* Participants must live in commuting distance from the hospital, as the training is organized as outpatient training
* Participants must be able to take instruction and master the Norwegian language

Exclusion Criteria:

* Patients who experience serious complications after surgery
* if a person has a disease that causes that one can not complete the planned training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Function1 | Pre-operative
  Function is evaluated using a questionnaire, Harris Hip Score (HHS) and by using 6-minute walk test (6MWT).
Function2 | Post-operative
  Function is evaluated using a questionnaire, Harris Hip Score (HHS) and by using 6-minute walk test (6MWT).
Funtion3 | After 12 weeks training
  Function is evaluated using a questionnaire, Harris Hip Score (HHS) and by using 6-minute walk test (6MWT).

SECONDARY OUTCOMES:
Muscle strength1 | Pre-operative
  Muscle strength around the operated hip are evaluated by measuring isometric muscle strength in hip-abduction and knee-extension using a hand-held dynamometer (HHD) from Lafayette Instruments.
Muscle strength2 | Post-operative
  Muscle strength around the operated hip are evaluated by measuring isometric muscle strength in hip-abduction and knee-extension using a hand-held dynamometer (HHD) from Lafayette Instruments.
Muscle strength3 | After 12 weeks training
  Muscle strength around the operated hip are evaluated by measuring isometric muscle strength in hip-abduction and knee-extension using a hand-held dynamometer (HHD) from Lafayette Instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Ottar Vasseljen, Principal Investigator — NTNU, Medisink fakultet, Institutt for samfunnsmedisin
Locations (1):
- St. Olavs Hospital, department Orkdal, Orkanger, Sør-Trøndelag, Norway